CLINICAL TRIAL: NCT04215016
Title: A Single-arm, Open-label, Dose Escalation Study to Explore Safety, Efficacy and Pharmacokinetics of Autologous Humanized Anti-CD19 and Anti-CD20 Dual Specific CAR-T Cells in Adult Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: Safety of Autologous Humanized Anti-CD19 and Anti-CD20 Dual Specific CAR-T Cells in Adult Patients With Diffuse Large B-cell Lymphoma
Acronym: A-02
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-19-05
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Relapsed or Refractory DLBCL Patients With Either CD19 or CD20 Positive
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Humanized anti-CD19 and anti-CD20 dual specific CAR-T cells (Experimental)
  Interventions: Biological: Autologous humanized anti-CD19 and anti-CD20 dual specific CAR-T Cells

INTERVENTIONS:
Biological: Autologous humanized anti-CD19 and anti-CD20 dual specific CAR-T Cells — Humanized anti-CD19 and CD20 bispecific autologous CAR-T cells injection: the first dose is 1.0×106 /kg, the second dose is 3.0×106 /kg, and the third dose is 8.0×106 /kg. Patients will receive lymphodepleting chemotherapy at least 1 week before CAR-T cell infusion.

SUMMARY:
This is a single-arm, open-label, dose escalation, phase I study, aiming to evaluate the safety and efficacy of Autologous Humanized Anti-CD19 and Anti-CD20 Dual Specific Chimeric Antigen Receptor (CAR) T-cells in patient with relapsed or refractory diffuse B cell lymphoma.

DETAILED DESCRIPTION:
CD19 CAR-T cell therapy has made breakthroughs in the treatment of B cell lymphoma and leukemia, but 30% of patients still have antigen escape, which may be related to variants in tumor cells and the expansion of CD19-negative tumor cells after treatment with CD19 CAR-T cells. CD19/CD20 bispecific CAR-T cell targeting multiple antigens can attack tumor cells while overcoming tumor antigen escape caused by a single target, maximizing efficacy and duration of treatment, and can also solve the problem of uneven distribution or low expression of single target on the tumor surface.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or her/his legally guardian(s) must sign the informed consent form approved by the Institutional Ethics Committee (IEC) prior to any screening procedures;
2. Subjects aged 18 years or older with relapsed or refractory DLBCL (primary mediastinal large B-cell lymphoma and transformed follicular lymphoma included), of which refractory is defined as:

   Have no response to the recent treatment including:
   * The best response to the treatment regimen is progressive disease (PD) ,or
   * stable disease (SD) which maintained less than 6 months after the last treatment, or
   * not suitable for autologous hematopoietic stem cell transplantation (ASCT), or ASCT refractory, including:

     * progressive disease after ASCT or relapse within 12 months (relapse must be confirmed by biopsy), or
     * If remedial treatment is given after ASCT, the subject must have no response or relapse after the last treatment.
3. Subjects who have previously received ≥2 lines treatment, and at least including:

   * Anti-CD20 monoclonal antibody(rituximab), unless the CD20 negative;
   * A chemotherapy regimen containing anthracyclines;
   * The DLBCL patients who transformed from follicular lymphoma must have previously received chemotherapy for follicular lymphoma and have developed chemotherapy-refractory diseases after transform to DLBCL.
4. Confirmation for either CD19 or CD20 positivity using immunohistochemistry or flow cytometry;
5. According to the initial evaluation, staging and response assessment of Hodgkin's and non-Hodgkin's lymphoma -the Lugano Classification (2014), there is at least one measurable lesion at baseline;
6. Life expectancy ≥12 weeks;
7. Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening;
8. Adequate organ function:

   Renal function defined as:
   * A serum creatinine of ≤1.5 × Upper Limit of Normal (ULN), or;
   * Estimated Glomerular Filtration Rate (eGFR) ≥60 ml/min/1.73m2；

   Liver function defined as:
   * ALT≤ 5 × Upper Limit of Normal (ULN) for age, and;
   * Total bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN.

   Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and blood oxygen saturation > 91% on room air;
9. Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA);
10. Adequate bone marrow reserve without transfusions defined as:

    * Absolute neutrophil count (ANC) >1×10^9 /L；
    * Absolute lymphocyte count (ALC) ≥0.3×10^9 /L；
    * Platelets ≥50×10^9 /L;
    * Hemoglobin > 8.0 g/dl;
11. Must have an apheresis product of non-mobilized cells or peripheral blood harvested cells accepted for manufacturing
12. Subjects who use the following drugs should meet the following criteria:

    * Steroids: Therapeutic doses of steroids must be stopped 2 weeks prior to A-02 infusion. However, the following physiological replacement doses of steroids are allowed: < 6 - 12 mg/m^2/day hydrocortisone or equivalent;
    * Immunosuppression: Any immunosuppressive medication must be stopped ≥ 4 weeks prior to sign the informed consent form;
    * Anti-proliferative therapy other than pretreatment chemotherapy within 2 weeks of A-02 infusion;
    * CD20 antibody-related treatment must be discontinued within 4 weeks of A-02 infusion or 5 half-lives (whichever is longer);
    * CNS disease prophylaxis must be stopped > 1 week prior to A-02 infusion (e.g. intrathecal methotrexate);
13. The investigator judged that the subject recovered from the toxicity of the previous anti-tumor treatment to grade 1 or below (except for special grade 2 or below toxicity that cannot be recovered in a short period of time, such as hair loss), suitable for pretreatment. Chemotherapy and treatment of CAR-T cells;
14. Women of child-bearing potential and all male subjects must agree to use highly effective methods of contraception for at least 12 months following A-02 infusion and until CAR-T cells are no longer present by PCR on two consecutive tests.

Exclusion Criteria:

1. Prior treatment with any cell therapy before signing the informed consent form, including CAR-T therapy;
2. Subjects with detectable cerebrospinal fluid malignant cells or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma;
3. Subjects with testicular invasion, including those who have had testicular resection;
4. Subjects with current or previous history of central nervous system disease, such as seizures, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system;
5. Subjects who have previously received allogeneic hematopoietic stem cell transplantation (HSCT); or suitable and consenting to Autologous hematopoietic stem cell transplantation (ASCT);
6. Chemotherapy other than lymphodepleting chemotherapy within 2 weeks of A-02 infusion;
7. Patients on oral anticoagulation therapy within 1 week of A-02 infusion;
8. Prior radiation therapy within 2 weeks of A-02 infusion;
9. Investigational medicinal product within the last 30 days prior to sign the informed consent form;
10. Subjects with active hepatitis B（defined as hepatitis B surface antigen positive, or hepatitis B core antibody positive with hepatitis B virus DNA detection value > 1000 copies/ml）or hepatitis C (HCV RNA positive)
11. Subjects positive for HIV antibody or treponema pallidum antibody;
12. Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to A-02 infusion)
13. Unstable angina and/or myocardial infarction within 6 months prior to sign the informed consent form;
14. Previous or concurrent malignancy with the following exceptions:

    * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to sign the informed consent form);
    * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to sign the informed consent form;
    * A primary malignancy which has been completely resected and in complete remission for ≥ 5 years;
15. Pregnant or nursing women (women of childbearing age were tested positive for pregnancy during screening period);
16. Cardiac arrhythmia not controlled with medical management;
17. Subjects with active neurological auto immune or inflammatory disorders (e.g. Guillain Barre Syndrome, Amyotrophic Lateral Sclerosis);
18. Other conditions that the investigator thinks he/she should not be included in this clinical trial, such as poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The types and Incidence of adverse events | Up to 12 months

SECONDARY OUTCOMES:
Overall response rate | Up to 12 months
  including CR and PR
Progression-free survival (PFS) | Up to 12 months
Response duration | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China